CLINICAL TRIAL: NCT07045259
Title: Effect of Exergaming Program Versus Neuromuscular Exercise on Locomotor and Cognitive Functions in Elderly People With Motor Cognitive Risk Syndrome
Brief Title: Effect of Exergaming Program Versus Neuromuscular Exercise in Elderly People With Motor Cognitive Risk Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulfidan Tokgoz, İstanbul Üniversitesi-Cerrahpasa, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/701
Record Dates: First submitted 2025-06-20; First posted 2025-07-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Motoric Cognitive Risk Syndrome; Elderly (People Aged 65 or More); Geriatric Patient; Exergaming; Neuromuscular Exercise
Keywords: Motoric Cognitive Risk Syndrome; Elderly; neuromuscular exercise; exergaming

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients who meet the inclusion criteria will be randomized into three treatment groups, structured exergaming and neuromuscular exercise training and control group with a 1:1 block allocation. Randomization will be performed by a researcher not involved in the study using a website (www.randomization.com). Interventions and assessments will be administered by physiotherapists. After the end of treatment, both groups will be re-evaluated using the same procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Neuromuscular Exercise Group (Active Comparator)
  Interventions: Other: Exergaming Exercise Training
- Exergaming Group (Active Comparator)
  Interventions: Other: The Neuromuscular Exercise Training program
- Control Group (No Intervention)

INTERVENTIONS:
Other: The Neuromuscular Exercise Training program — The Neuromuscular Exercise Training program will be carried out in groups of 2 people for 45 minutes/2 days/8 weeks. The exercise program will consist of warm-up, loading and cooling phases. The warm-up phase will consist of flexibility exercises, mini squat and roll down etc. exercises to prepare the individual for exercise. The loading phase will consist of a cognitive-based neuromuscular exercise program aiming to provide stabilization, increase in balance, neuroplasticity and motor control and is planned to include strengthening exercises, stabilization exercises, balance-proprioceptive exercises and neuromuscular control exercise training with visual feedback. The exercises will progress gradually from easy to difficult with increasing repetition and set numbers.
  Arms: Exergaming Group
Other: Exergaming Exercise Training — In our study, Xbox One Kinect game console and Kinect sensor will be used within the scope of Exergaming. Exergaming program will be carried out in groups of 2 people for 45 minutes/ 2 days/ 8 weeks. It will consist of warm-up, loading and cooling phases. The games to be used for the Exergaming program were selected from games that include locomotor and cognitive repetitive tasks. The selected exergames involve repetitive locomotor and cognitive tasks. Piano step will be utilized during the warm-up for its rhythm-based movement patterns. For the conditioning phase, lower extremity exercises will include Reflex Ridge, River Rush, and Rallyball (Kinect Adventures), while upper extremity exercises will consist of Bowling, Table Tennis, Swimming (Kinect Sports), and Fruit Ninja. A progressive training approach will be followed, with game difficulty levels increasing incrementally as the sessions advance.
  Arms: The Neuromuscular Exercise Group

SUMMARY:
The primary aim of our study is to compare the effects of neuromuscular exercise training versus structured exergaming program on locomotor and cognitive functions in elderly individuals with Motor Cognitive Risk (MCR), which defines the transition state between typical aging and dementia and mild cognitive impairment. This study aims to present for the first time the effects of neuromuscular exercise training and exergaming program on locomotor and cognitive functions in elderly individuals with MCR with comparative results.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years of age
* Having a Barthel Daily Living Activities Index score of ≥ 90
* Having a Mini Mental Status Score (MMSE) of ≥24
* Having the ability to walk with or without a walking aid
* Having a slow walking speed
* Having subjective memory complaints

Exclusion Criteria:

* Presence of Dementia
* Major Depression
* Generalized Anxiety Disorder and Delirium
* Parkinson's Disease
* Anemia
* Thyroid Disease
* Vitamin B12 Deficiency
* Malnutrition
* Terminal Illness
* Hearing or Visual Impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG) | From enrollment to the end of treatment at 8 weeks
  TUG test is a frequently used field test to evaluate mobility, balance, fall risk and walking in elderly individuals (Magda,2024; (Racha, 2023). The test involves the individual getting up from a chair, walking 3 meters, turning, and sitting. The time taken to complete this series of movements is measured and recorded using a stopwatch (Racha, 2023).
Stair Climbing Test (SCT) | From enrollment to the end of treatment at 8 weeks
  The stair climbing test is frequently used in the evaluation of locomotor functions in elderly individuals. The validity and reliability of the STAIR, which has been investigated in elderly people with knee osteoarthritis, has been reported to have a test-retest reliability coefficient of 0.93 and high reliability (Jose, 2021). In our study, they will be asked to ascend and descend 4 steps, each of which is 50 cm wide, 15 cm high and 25 cm deep, as quickly but safely as possible. They will be able to use the handrails when they need to while ascending or descending the stairs, and the total time taken to complete the task will be measured in seconds with a stopwatch.
Cognitive Officer TUG-SCT | From enrollment to the end of treatment at 8 weeks
  In our research
  * Counting backwards from 50 by threes
  * Cognitive officer TUG and SCT tests will be conducted to answer the questions prepared by the researchers as yes if red and no if blue, and the results will be recorded in terms of time (Li, 2023).

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | From enrollment to the end of treatment at 8 weeks
  Short Physical Performance Battery (SPPB) is a field test designed to evaluate the physical performance of elderly people, helps interpret their functional abilities, and gives an idea about the individual's biological age (Pavasini, 2016). SPPB, which is frequently used in elderly individuals in the literature, consists of the categories of static balance, 4-meter walking test, and 5-times sit-to-stand test (Corsonello, 2012 ). The balance test in SPPB includes three different postures: side-by-side, semi-tandem, and tandem. Each posture is held for up to 10 seconds. The ability to maintain these positions gives an idea about the individual's balance abilities (Cisternas, 2024). It is emphasized in the literature that the balance test, together with other components of SPPB, can predict all-cause mortality (Pahor, 2014). In our research, SPPB will be used to evaluate the static balance ability, walking speed, functional capacity,
Dynamic Gait Index (DGI) | From enrollment to the end of treatment at 8 weeks
  The Dynamic Gait Index (DGI) is a widely accepted functional gait tool for assessing the risk of falls and functional stability while walking in the elderly (Shumway-Cook et al., 2013). In the literature, DGI is used as a valid, reliable, cheap and fast tool to assess the gait and balance of elderly individuals (Alghwiri, 2014). It consists of eight items including normal walking on level ground, walking with speed changes, walking with horizontal head movements, walking with vertical head movements, walking with pivot turns, walking by jumping over obstacles, taking steps around obstacles and climbing up and down stairs. Each item is rated on a 4-point scale ranging from 0 (severe impairment) to 3 (independent walking). The maximum total score can be 24. The scale, whose validity and reliability in Turkish in elderly individuals was conducted by Zirek, will be used to comprehensively assess walking in our study (Zirek, 2023).
Reaction speed assessment | From enrollment to the end of treatment at 8 weeks
  Reaction speed is defined as the duration between the stimulus reaching the central nervous system and the execution of the appropriate motor response. It is closely associated with cognitive functions such as attention, processing speed, motor planning, and executive functions. Considering the age-related decline in processing speed and motor response, the Light Trainer Flash Light Exercise System (Reaction X) will be utilized to evaluate these parameters.
  Upper Limb Reaction Speed Assessment
  The assessment consists of two protocols, each lasting 30 seconds:
  Choice Reaction (Colored Light): To evaluate decision-making and reasoning, participants must respond to color-coded stimuli (e.g., blue light for the right hand and red light for the left).
  Lower Limb Reaction Speed Assessment This protocol evaluates decision-making and balance concurrently. Using their dominant leg, participants will deactivate specific colored sensors for 30 seconds.
Performance-Oriented Mobility Assessment | From enrollment to the end of treatment at 8 weeks
  The Performance-Oriented Mobility Assessment (POMA), introduced to the literature by Tinetti in 1986, is frequently used to assess balance and gait in elderly individuals and to assess the risk of falls in individuals with conditions affecting balance and gait (Tinetti, 1986). POMA, whose Turkish validity and reliability were conducted by Ağırcan, will be used in our research for the comprehensive assessment of gait and balance (Ağırcan, 2009). Permissions from the authors are provided as an attachment.
Berg Balance Assessment | From enrollment to the end of treatment at 8 weeks
  Berg Balance Test (BBS), one of the frequently used tests in balance assessment in elderly individuals, has a test-retest reliability with an ICC (Intraclass Correlation Coefficient) of 0.91 and high inter-rater reliability with an ICC of 0.97 (Neuls, 2011). BBS, which consists of 14 different tasks or activities, is scored from 0 to 4 for tasks such as sitting to standing, standing without support, sitting without support, etc. The total score varies between 0 and 56, with a high score being interpreted as better balance. The scale, which was validated in Turkish by Şahin and colleagues, shows a high risk of falling, a score of 0 to 20 indicates a moderate risk of falling, a score of 21 to 40 indicates a moderate risk of falling, and a score of 41 to 56 indicates a low risk of falling (Sahin, 2008).
Physical Activity Enjoyment Scale | From enrollment to the end of treatment at 8 weeks
  The Physical Activity Enjoyment Scale is one of the scales used to measure enjoyment in physical activity. The test-retest reliability of the scale was reported to be 0.69, showing strong internal consistency and reliability (Weyland et al., 2024). The Turkish validity and reliability of the scale, which consists of 8 items and a single dimension, was conducted by Özkurt et al. in 2022, and it was reported that the Turkish form can be used as a valid and reliable measurement tool (Özkurt, 2022).
Exercise Adherence and Participation Rate | From enrollment to the end of treatment at 8 weeks
  To monitor exercise adherence, session attendance will be recorded by the researchers using an Exercise Program Attendance Tracking Chart. Participants who fail to attend four or more sessions (representing a dropout/non-attendance rate of ≥25%) of the 16-session program will be excluded from the study. Furthermore, adherence rates will be compared across the exercise groups.

OTHER OUTCOMES:
Satisfaction Level | From enrollment to the end of treatment at 8 weeks
  Participant satisfaction levels regarding the program will be evaluated using a researcher-developed questionnaire. Participants will be asked to rate their overall satisfaction with the intervention, their willingness to participate in the program again if it were repeated, and other satisfaction-related metrics on a 10-point scale (ranging from 1 to 10, where 10 represents the highest level of satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Gulfidan TOKGÖZ, Lecturer, PhD (c), Principal Investigator — İstanbul University-Cerrahpasa; Saime Nilay ARMAN, Assoc. Prof. Dr., Study Director — İstanbul University-Cerrahpasa
Locations (1):
- Balıkesir Üniversitesi, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davranche K, Burle B, Audiffren M, Hasbroucq T. Physical exercise facilitates motor processes in simple reaction time performance: an electromyographic analysis. Neurosci Lett. 2006 Mar 20;396(1):54-6. doi: 10.1016/j.neulet.2005.11.008. Epub 2006 Jan 10. PMID 16406344
- [Background] Garcia MAC, Souza VH. The (un)standardized use of handheld dynamometers on the evaluation of muscle force output. Braz J Phys Ther. 2020 Jan-Feb;24(1):88-89. doi: 10.1016/j.bjpt.2019.10.004. Epub 2019 Nov 13. No abstract available. PMID 31740163
- [Background] Zirek E, Mustafaoglu R, Cicek A, Ahmed I, Mavromoustakos S. Reliability and Validity of the Turkish Version of the Modified Dynamic Gait Index in the Elderly. Eval Health Prof. 2023 Jun;46(2):135-139. doi: 10.1177/01632787221128311. Epub 2022 Sep 17. PMID 36121068
- [Background] Alghwiri AA. Reliability and validity of the Arabic Dynamic Gait Index in people poststroke. Top Stroke Rehabil. 2014 Mar-Apr;21(2):173-9. doi: 10.1310/tsr2102-173. PMID 24710977
- [Background] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Background] Corsonello A, Lattanzio F, Pedone C, Garasto S, Laino I, Bustacchini S, Pranno L, Mazzei B, Passarino G, Incalzi RA; Pharmacosurveillance In The Elderly Care Pvc Study Investigators. Prognostic significance of the short physical performance battery in older patients discharged from acute care hospitals. Rejuvenation Res. 2012 Feb;15(1):41-8. doi: 10.1089/rej.2011.1215. Epub 2011 Oct 17. PMID 22004280
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Li Y, Yu N, Zhang C, Song Q, Wang J, Sun W. Test-retest reliability of kinematic and kinetic parameters during dual-task stair walking in the elderly. Front Physiol. 2023 May 9;14:1177159. doi: 10.3389/fphys.2023.1177159. eCollection 2023. PMID 37228826
- [Background] Casana J, Calatayud J, Silvestre A, Sanchez-Frutos J, Andersen LL, Jakobsen MD, Ezzatvar Y, Alakhdar Y. Knee Extensor Muscle Strength Is More Important Than Postural Balance for Stair-Climbing Ability in Elderly Patients with Severe Knee Osteoarthritis. Int J Environ Res Public Health. 2021 Mar 31;18(7):3637. doi: 10.3390/ijerph18073637. PMID 33807414
- [Background] Soubra R, Mourad-Chehade F, Chkeir A. Automation of the Timed Up and Go Test Using a Doppler Radar System for Gait and Balance Analysis in Elderly People. J Healthc Eng. 2023 Jun 29;2023:2016262. doi: 10.1155/2023/2016262. eCollection 2023. PMID 37426725
- [Background] Reis M, Teixeira M, Carvao C, Martins AC. Validity and Reliability of the Self-Administered Timed Up and Go Test in Assessing Fall Risk in Community-Dwelling Older Adults. Geriatrics (Basel). 2025 Apr 29;10(3):62. doi: 10.3390/geriatrics10030062. PMID 40407569